CLINICAL TRIAL: NCT06553079
Title: Development of the Surgeon Satisfaction Self-Assessment Questionnaire for Shoulder Arthroscopy
Status: Not yet recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, İnci Hazal Ayas, Principal Investigator, Gazi University
Other Study IDs: Iayas11
Record Dates: First submitted 2024-08-10; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Surgeon Satisfaction; Shoulder Arthroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgeons Performing Shoulder Arthroscopy: This is the main group of interest and includes surgeons who regularly perform shoulder arthroscopy. They will be the primary respondents to the survey and will provide insights into the factors affecting their surgical satisfaction.
  Interventions: Other: Surgeon Satisfaction Self-Assessment Questionnaire for Shoulder Arthroscopy

INTERVENTIONS:
Other: Surgeon Satisfaction Self-Assessment Questionnaire for Shoulder Arthroscopy — The intervention in this study involves the administration of the "Surgeon Satisfaction Self-Assessment Questionnaire for Shoulder Arthroscopy," a newly developed tool designed to measure various aspects of surgeon satisfaction related to shoulder arthroscopy procedures.

SUMMARY:
This observational study aims to develop and validate the "Surgeon Satisfaction Self-Assessment Questionnaire for Shoulder Arthroscopy." The study involves conducting in-depth interviews with surgeons who perform shoulder arthroscopy to identify key factors influencing their surgical satisfaction, including individual, patient-related, and surgical equipment-related factors. Based on the insights gained from these interviews, a comprehensive questionnaire will be developed. The questionnaire will then undergo validation processes, including assessments of content, construct, criterion, and reliability, to ensure it accurately and consistently measures surgeon satisfaction. The final validated tool is intended to provide a reliable method for surgeons to self-assess their satisfaction with shoulder arthroscopy procedures, contributing to improved surgical practices and outcomes.

DETAILED DESCRIPTION:
The "Surgeon Satisfaction Self-Assessment Questionnaire for Shoulder Arthroscopy" is being developed to address the need for a standardized tool to evaluate surgeon satisfaction in the context of shoulder arthroscopy. This study is structured into two primary phases: survey development and validation.

Phase 1: Survey Development In the initial phase, semi-structured interviews will be conducted with a diverse group of surgeons who specialize in shoulder arthroscopy. These interviews will explore various dimensions of surgical satisfaction, including technical factors, patient outcomes, surgical equipment performance, and team dynamics. The qualitative data obtained from these interviews will be analyzed to identify recurring themes and factors that are crucial to surgeon satisfaction. Based on these findings, a draft questionnaire will be developed, ensuring that it comprehensively covers all relevant aspects of the surgical experience.

Phase 2: Validation Process Once the questionnaire is drafted, it will undergo a rigorous validation process. Content validity will be established by consulting with a panel of experts in orthopedic surgery and psychometrics to ensure that the questionnaire items are both relevant and exhaustive. Construct validity will be tested using factor analysis to determine the underlying structure of the questionnaire and to ensure it accurately measures the intended constructs of satisfaction. Criterion validity will be assessed by comparing the questionnaire outcomes with established benchmarks or other validated tools. Additionally, the questionnaire's reliability will be evaluated through test-retest and internal consistency measures Cronbach's alpha.

ELIGIBILITY:
Inclusion Criteria:

* Orthopedic Surgeons:Must be a licensed orthopedic surgeon actively performing shoulder arthroscopy procedures.
* Participants must be willing to provide informed consent and participate in both the questionnaire development (including interviews) and the validation phases of the study.
* Participants must be proficient in the language in which the questionnaire is administered to ensure accurate and meaningful responses.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of orthopedic surgeons who specialize in shoulder arthroscopy and are actively engaged in performing these procedures. Participants will be recruited from a variety of clinical settings, including academic medical centers, private practices, and specialized orthopedic clinics. The surgeons included in the study will have diverse levels of experience, ranging from early-career surgeons with low practice to highly experienced surgeons with decades of experience in the field.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Validation of the Surgeon Satisfaction Self-Assessment Questionnaire for Shoulder Arthroscopy | 6 months
  The primary outcome measure is the successful development and psychometric validation of the Surgeon Satisfaction Self-Assessment Questionnaire for Shoulder Arthroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Ulunay Kanatlı, Professor, Study Director — Gazi University
Locations (1):
- Gazi University Hospital, Ankara, Turkey (Türkiye)